CLINICAL TRIAL: NCT02638467
Title: Allogeneic Haematopoietic Stem Cell Transplantation From a Matched Donor in Patients With Chronic Myeloid Leukemia Failing to Gain Normal Hemopoiesis Under TKIs Therapy
Brief Title: Allogeneic Stem Cell Transplantation in Chronic Myeloid Leukemia Failing TKIs Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Milano Bicocca (Other)
Collaborators: IRCCS San Raffaele (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: alloCML
Record Dates: First submitted 2015-12-09; First posted 2015-12-23 (Estimated); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: Leukemia; Myelogenous; Chronic; BCR-ABL Positive
MeSH Terms: conditions — Leukemia; Bronchiolitis Obliterans Syndrome | interventions — bosutinib; Bone Marrow Transplantation; SLC25A33 protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bosutinib and Bone Marrow Transplant (Experimental): Subjects will receive 400mg of bosutinib from day at least -45 to day -15 to assess the sensitivity of patient Chronic Myeloid Leukemia (CML) to this TKI. Patients will be transplanted with the aim to transplant > 3 x 106 CD34+ cells/kg Body Weight (BW) recipient from bone marrow or > 3 x 108 nucleated cells/kg BW recipient from bone marrow. Then, subjects will receive 400mg of bosutinib once daily from day +30 after transplant.
  Interventions: Drug: Bosutinib; Procedure: Bone Marrow Transplant; Drug: Bone Marrow cells

INTERVENTIONS:
Drug: Bosutinib — Subjects will receive 400mg of bosutinib once daily from day +30 after transplant, by mouth with food, preferably in the morning. Bosutinib will also be administered from day at least -45 to day -15 to assess the sensitivity of patient CML to this TKI.
  Other Names: Bosulif; SKI-606
Procedure: Bone Marrow Transplant — Samples of the unrelated stem cell graft shall be characterised with respect to the number of CD34 positive cells per kg body weight of the recipient.
  The number of transplanted CD34 positive cells per kg body weight (BW) of the recipient shall be recorded in the Case Report Form (CRF). If the transplant was cryopreserved the number of viable CD34 positive cells has to be determined after thawing and documented.
  The goal is to transplant > 3 x 106 CD34+ cells/kg BW recipient from bone marrow or > 3 x 108 nucleated cells/kg BW recipient from bone marrow
Drug: Bone Marrow cells

SUMMARY:
Patients newly diagnosed with chronic phase chronic myeloid leukemia undergo treatment with TK inhibitors (TKI). A possible cause of TK failure is represented by the insufficient recovery of normal Ph- hematopoiesis during TKI treatment, with consequent severe cytopenias that limit TKI adequate administration. Although rare, this event happens in a proportion of 4-5% of CML patients. Our hypothesis is to circumvent this peculiar condition by providing a normal hematopoiesis from a HLA-matched donor (Human Leukocyte Antigen). The transplant procedure is therefore intended in providing a sustained hematopoiesis that will allow an early treatment with an adequate dosing of TKI. The transplant procedure planned in our study is built on all available evidences to provide the lowest incidence of acute and chronic GvHD (Graft-versus-host disease). Therefore, a bone marrow will be the preferential source and a GvHD prophylaxis based on Anti-thrombocyte globulin (ATG) and Cyclosporine/Methotrexate will be used according to standard current experience in the field of family and unrelated donors. The pre-transplant TKI will be continued until aplasia will develop, in order to decrease the tumor load as much as possible.The use of TKIs shortly after transplant carries the risk of inhibiting the newly transplanted hematopoietic cells, as Kit, an important kinase in normal bone marrow cells, is frequently blocked by Abl inhibitors. The use of bosutinib as post-transplant therapy is justified by the lack of Kit inhibition that distinguishes bosutinib from all other TKIs, and which could allow a minimal inhibitory activity against the transplanted normal bone marrow.

ELIGIBILITY:
Inclusion Criteria:

1. Chronic Myeloid Leukaemia -CML- in chronic phase (CP)
2. Failure to achieve at least a Major Cytogenetic Response (MCyR) after a minimum of 18 months of TKIs treatment
3. Inability to tolerate 3 months of uninterrupted full dose TKIs therapy due to hematological toxicity
4. A minimum of three treatment interruptions due to hematological toxicity Availability of a HLA-identical related donor (Matched Related Donor, MRD)
5. Availability of unrelated donor (Matched Unrelated Donor, MUD) satisfying the criteria of a 10/10 antigen match at (Human Leukocyte Antigen) HLA-A, -B, -C and - DRB1, -DQB1 at high resolution typing, or 9/10 with a permissive - DP disparity according to Fleischhauer model (Crocchiolo et al, Blood 2009)
6. Target graft size (bone marrow):
7. bone marrow: > 3 x 106 CD34+ cells/kg BW recipient or > 3 x 108 nucleated cells/kg BW
8. Karnofsky Index > 80 %
9. Age ≥18 and ≤70 years
10. Adequate contraception in female patients of child-bearing potential
11. Written informed consent

Exclusion Criteria:

1. Secondary malignancies
2. A hematopoietic cell transplantation-specific comorbidity index (Sorror et al Appendix C) > 4
3. Known and manifested malignant involvement of the Central Nervous System (CNS)
4. Active infectious disease
5. Active human immunodeficiency virus (HIV), Hepatitis B virus (HBV) or Hepatitis B virus (HCV) infection
6. Impaired liver function (Bilirubin > upper normal limit; Transaminases > 3.0 x upper normal limit)
7. Impaired renal function (Creatinine-clearance < 60 ml/min; Serum Creatinine > 1.5 x upper normal limit).
8. Pleural effusion or ascites > 1.0 L
9. Pregnancy or lactation
10. Known hypersensitivity to Busilvex and/or fludarabine 11 Non-co-operative behaviour or non-compliance 12 Psychiatric diseases or conditions that might impair the ability to give informed consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2018-11-29 (Actual); Study Completion 2020-02 (Actual)

PRIMARY OUTCOMES:
Efficacy as assessed by the percentage of patients with Complete Cytogenetic Response (CCyR) | 12 months
  The percentage of patients with Complete Cytogenetic Response (CCyR) will be calculated as the complement to the percentage of failures on the total number of patients treated, where failure includes the following events: no engraftment, death within 12 months, no CCyR at 12 months.

SECONDARY OUTCOMES:
Overall Survival | 12 months
Percentage of patients with engraftment | 12 months
percentage of patients with complete chimerism (95%) | Day +28, +56 and +100
Evaluation of Major Cytogenetic Response (MCyR) | 12 months
  Major Cytogenetic Response (MCyR) is < 36% Ph+ metaphases
Evaluation of molecular responses | 12 months
  Molecular response is defined
  * Complete: if there is undetectable BCR-ABL transcript
  * Major: if ratio BCR/ABL <= 0.1% on International Scale
Relapse incidence (RI) | 12 months
Incidence of non-relapse mortality (NRM) | Within day +28 and +360
Incidence and severity of acute and chronic graft vs. host disease (GvHD) | 12 months
Quality of Life (QoL) | 12 months
  Evaluation of QoL with EQ-5D-5L (Italian - Version 2) and FACT-Leu (Italian -Version 4)
Overall Survival (OS) | 36 months
  2 years after transplantation of the last patient included (this is intended to allow evaluations of all expected major molecular responses)
Progression Free Survival (PFS) | 36 months
  2 years after transplantation of the last patient included (this is intended to allow evaluations of all expected major molecular responses)
Relapse Incidence (RI) | 36 months
  2 years after transplantation of the last patient included (this is intended to allow evaluations of all expected major molecular responses)
Chronic Graft-versus-host Disease (cGvHD) | 36 months
  2 years after transplantation of the last patient included (this is intended to allow evaluations of all expected major molecular responses)

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Gambacorti-Passerini, MD, Principal Investigator — University of Milano Bicocca
Locations (2):
- Italy (2):
  - ASST-Monza, Monza, Italy/MB
  - Ospedale San Raffaele, Milan, MI

REFERENCES:
- [Background] Redaelli A, Bell C, Casagrande J, Stephens J, Botteman M, Laskin B, Pashos C. Clinical and epidemiologic burden of chronic myelogenous leukemia. Expert Rev Anticancer Ther. 2004 Feb;4(1):85-96. doi: 10.1586/14737140.4.1.85. PMID 14748660
- [Background] Heisterkamp N, Stephenson JR, Groffen J, Hansen PF, de Klein A, Bartram CR, Grosveld G. Localization of the c-ab1 oncogene adjacent to a translocation break point in chronic myelocytic leukaemia. Nature. 1983 Nov 17-23;306(5940):239-42. doi: 10.1038/306239a0. PMID 6316147
- See also: Cancer Facts and Figures. 2006, American Cancer Society — http://www.cancer.org